CLINICAL TRIAL: NCT05069987
Title: Anxiety Reduction in TAVI Using Virtual Reality Trial
Acronym: ART-VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Prof. Dr. Nicolas Van Mieghem, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2021-0417; NL77298.078.21 (Other: Central Commissie Mensgebonden Onderzoek)
Record Dates: First submitted 2021-09-20; First posted 2021-10-06 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Aortic Stenosis, Severe; Anxiety
Keywords: Immersive Virtual Reality; Procedural Anxiety; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis; Anxiety Disorders | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned, in a 1:1 ratio, to either procedural VR-immersion or non-VR control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-immersion (Experimental)
  Interventions: Other: Virtual Reality Immersion
- Non-VR control (No Intervention)

INTERVENTIONS:
Other: Virtual Reality Immersion — An immersive virtual reality experience will be generated by a head mounted device which shows the user pre-recorded videos (SynVR Relax & Distract, SyncVR Medical BV, Utrecht, The Netherlands). These videos are recorded in 360 degree views and matched with the users' viewing direction by the head mounted device matches. The user will not be able to see its in vivo surroundings (i.e. the Cathlab) and will be focused on the digital content. The VR immersion will be put into place throughout the entire TAVR procedure starting before femoral access obtainment and ending after access closure.
  Arms: VR-immersion

SUMMARY:
The ART-VR Trial is an international multi-center, open label, randomized controlled trial evaluating the effect of an immersive VR environment on procedural anxiety in patients undergoing transfemoral aortic valve replacement (TAVR) under local anaesthesia.

DETAILED DESCRIPTION:
Virtual reality (VR) allows patients to be fully immerged in an engaging, interactive 3D environment. Its applications are broad and include treatment of phobias, stress-disorders, pain reduction. Recently, VR has been adopted in various medical procedures to reduce pre- and per-procedural anxiety. In TAVR, per-procedural VR immersion could potentially reduce patient anxiety leading to increased overall patient satisfaction. However, contemporary large scale, randomized evidence on VR application in TAVR is lacking.

The objective of this trial is to evaluate the effect of an immersive VR environment on procedural anxiety in patients undergoing TAVR under local anaesthesia in a randomized controlled setting. A total of 150 patients with severe aortic stenosis (AS) who undergo transfemoral TAVR under local aneasthesia will be included. The main study endpoint is procedural anxiety assessed on a visual analogue scale (VAS) directly post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptomatic severe aortic stenosis
* Indication for transfemoral TAVI under local anaesthesia per local heart team consensus
* Patient is able to understand and sign written informed consent
* Patient speaks Dutch, German or English

Exclusion Criteria:

* Need for emergent TAVI
* Need for planned concomitant cardiac intervention during index procedure
* History of TAVI under local anesthesia/conscious sedation
* Chronic use of benzodiapines, opioids, pregabalin or antidepressants
* History of opioid use (within 8-30 days prior to randomization)
* Claustrophobia
* Any psychiatric illness diagnosed by a psychiatrist or psychologist
* Blindness or severe visual impairment despite visual aid (glasses, contact lenses)
* Epilepsy
* Extensive cognitive impairment (MMSE <21 or as diagnosed by geriatrician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Procedural Anxiety | Immediately after the TAVR procedure
  Procedural anxiety assessed on a visual analogue scale directly post-procedure. Range: 0 (no anxiety) to 10 (worst anxiety).

SECONDARY OUTCOMES:
Change of Anxiety | 1 day (From directly before the TAVR procedure until directly after the TAVR procedure)
  Difference between pre-procedural and post-procedural anxiety visual analogue scale scores
Procedural Pain | Immediately after the TAVR procedure
  Procedural pain assessed on a visual analogue scale directly post-procedure. Range: 0 (no pain) to 10 (worst pain).
Procedural Use of Sedatives | Up to 1 day (Depending on procedure duration)
  Procedural sedative use and dosage. Amount of benzodiazepine used in milligrams
Procedural Use of Analgesics | Up to 1 day (Depending on procedure duration)
  Procedural analgesic use and dosage. Amount of Lidocaine (or equivalent) used in milligrams
Patient Procedural Satisfaction | One day post procedure
  Procedural satisfaction assessed after 24hrs using for procedures under regional anaesthesia. Score assessed on a visual analogue scale. Range: 0 (not at all satisfied) to 10 (very satisfied).

OTHER OUTCOMES:
Patient reported procedural Nausea and Vomiting | Up to 1 day (Depending on procedure duration)
  Patient reported nausea and vomiting during the procedure (yes/no)
Admission time | Up to 7 days
  Time leaving cathlab until discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol